CLINICAL TRIAL: NCT05113875
Title: Health System Dynamic & Resource Requirement in a South African COVID-19 Field
Brief Title: Health System Dynamic & Resource Requirement in a South African COVID-19 Field Hospital
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Ruth Verity Passchier, Doctor, University of Cape Town
Other Study IDs: African Covid19 Field Hospital
Record Dates: First submitted 2021-11-03; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Field Hospitals; COVID-19 Pandemic; Health Systems; Global Health; Health Resources; Low-Income Population
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Patients: Completed Sample of all patients admitted to the Mitchells Plain Hospital of Hope COVID-19 Field Hospital between January 1st and February 29th 2021. All patients were diagnosed with COVID-19 prior to admission to the hospital and were transferred directly from a referring hospital.

SUMMARY:
The aim of this study is to describe the patient clinical profile, resource requirements, and health system dynamics in a field hospital during the second wave of the Coronavirus (COVID-19) pandemic, leading to the outbreak of viral severe acute respiratory syndrome (SARS-CoV-2 virus), in South Africa. By describing the field hospital in this unique setting, the investigators hope to provide an efficient guide to similar settings across low- and middle-income countries.

This was a retrospective, single-center study. A total of 596 patients with confirmed COVID-19 were admitted to Mitchells Plain Hospital of Hope (MPHOH), Cape Town, South Africa, between January 1st and February 28th, 2021. Patient clinical characteristics, outcome, and resource allocation was collected. Daily hospital dynamics, including admissions, discharges, deaths and oxygen use was analyzed and compared to the local and national COVID-19 incidence rates.

DETAILED DESCRIPTION:
The aim of the study is to amplify what is known about field hospitals in resource-constrained setting, so as to guide meaningfully the future COVID-19 public health response. Understanding not only the patient profile, but clinical resource requirements, and health system dynamic in a South African field hospital during the second wave of the COVID-19 pandemic can help in preparation for a future infection surge. This will shed light on the extent and timing of excess demand for intermediate care facilities for COVID-19 during peak infection periods in this region. Furthermore, lessons learnt here can guide efforts in similar settings across low-and middle-income countries.

Data was collected on all patients admitted to MPHOH between January 1st and February 28th 2021 using notes from patient folders' and an electronic hospital records systems. Patient demographics, clinical profile, resource utilization; as well as the hospital dynamics were collected. COVID-19 incidence rates were collected from the National Institute for Infectious Diseases, South Africa

A descriptive data analysis was performed to report the number, mean, median, and range of all relevant values. Hospital level data were summarized into weekly intervals, described and compared to COVID-19 incidence rates. Statistical data analysis was performed using R Statistical Computing program and Microsoft Excel.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Mitchells Plain Hospital of Hope COVID-19 field hospital between 1st January 2021 and 29th February 2021. Patients admitted to the hospital must have been: over 18years of age, diagnosed with COVID-19 via polymerase chain reaction (PCR) test, transferred from a referring facility.

Exclusion Criteria:

* No patients were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is from an underserved community utilizing public health services. The population in based in Mitchells Plain, Cape Town South Africa.
Sampling Method: Non-Probability Sample
Enrollment: 596 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Patient Demographics | January 1st to February 29th 2021
  Patient age (in numbers)
Patient Demographics | January 1st to February 29th 2021
  Patient sex (male or female)
Patient Clinical Condition | January 1st to February 29th 2021
  Patient medical comorbidities on admission (categorical)
Patient Clinical Condition | January 1st to February 29th 2021
  If patient diabetic, type of diabetic treatment received in hospital (oral vs insulin therapy)
Patient Clinical Condition | January 1st to February 29th 2021
  If patient diabetic, glycated haemoglobin (HBA1C) level during admission (in numbers)
Patient Clinical Condition | January 1st to February 29th 2021
  Patient clinical complications during hospital admission (categorical)
Patient Clinical Condition | January 1st to February 29th 2021
  If patient received antibiotic treatment during admission, name of infection treated (categorical)
Patient Clinical condition | January 1st to February 29th 2021
  Patient ICU priority triage score on admission (in numbers)
Hospital Human Resources Utilized | January 1st to February 29th 2021
  Number of patients who utilized palliative care services (in numbers)
Hospital Human Resources Utilized | January 1st to February 29th 2021
  Number of patients who utilized dietician services (in numbers)
Hospital Human Resources Utilized | January 1st to February 29th 2021
  Number of patients who utilized physiotherapy services (in numbers)
Hospital Physical Resources Utilized | January 1st to February 29th 2021
  Number of patients requiring oxygen therapy during admission (in numbers)
Hospital Physical Resources Utilized | January 1st to February 29th 2021
  Type of oxygen therapy utilized by each patient (Categorical: nasal prong oxygen; face mask oxygen; or high flow oxygen)
Hospital Physical Resources Utilized | January 1st to February 29th 2021
  Duration of oxygen therapy for each patient (in days)
Hospital Physical Resources Utilized | January 1st to February 29th 2021
  Number of patients requiring antibiotic treatment (in numbers)
Hospital Physical Resources Utilized | January 1st to February 29th 2021
  If patient required antibiotic therapy, name of antibiotic given (categorical)
Hospital Physical resources Utilized | January 1st to February 29th 2021
  Patient duration of hospital stay (in days)
Health System Dynamics | January 1st to February 29th 2021
  Daily number of patients admitted to hospital (in numbers/day)
Health System Dynamics | January 1st to February 29th 2021
  Daily number of inpatients at hospital (in numbers/day)
Health System Dynamics | January 1st to February 29th 2021
  Daily number of patients discharged from hospital (in numbers/day)
Health System Dynamics | January 1st to February 29th 2021
  Daily number of patient deaths (in numbers/day)
Health System Dynamics | January 1st to February 29th 2021
  Daily number of patients transferred out of hospital to another medical facility (in numbers/day)
Health System Dynamics | January 1st to February 29th 2021
  Daily hospital bed capacity (in numbers/day)
Health System Dynamics | January 1st to February 29th 2021
  Daily hospital oxygen consumption (in kg/day)
Health System Dynamics | January 1st to February 29th 2021
  Name of hospital from which each patient was referred from (categorical)
Local Incidence rates of COVID-19 infections | December 1st 2020 to February 29th 2021
  South African National COVID-19 incidence rates per week (in numbers/week)
Local Incidence rates of COVID-19 infections | December 1st 2020 to February 29th 2021
  Western Cape Provincial COVID-19 incidence rates per week (in numbers/week)

CONTACTS AND LOCATIONS:
Locations (1):
- Mitchells Plain Hospital of Hope Covid-19 Field Hospital, Lentegeur Hospital, Cape Town, Western Province, South Africa

IPD SHARING:
Plan to Share IPD: No
Individual participant data and hospital level data will be available to the public on completion of the research